CLINICAL TRIAL: NCT07105202
Title: Shorter Weaning From Invasive Ventilation With Levosimendan: a Randomized, Double-blind, Multicentre Study in Critically Ill Patients
Brief Title: Shorter Weaning From Invasive Ventilation With Levosimendan
Acronym: WEANLESS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-518810-23-00; 2024-518810-23-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-09; First posted 2025-08-05 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-05

CONDITIONS: Mechanical Ventilation; Weaning Failure
Keywords: mechanical ventilation; weaning; critically ill patients; levosimendan; diaphragm
MeSH Terms: interventions — Simendan; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): Participants randomized to this arm will receive intravenous levosimendan. This group will consist of 125 patients.
  Interventions: Drug: levosimendan; Other: Standard care
- Control group (Placebo Comparator): Participants randomized to this arm will receive a placebo consisting of Soluvit. This group will consist of 125 participants.
  Interventions: Drug: Soluvit; Other: Standard care

INTERVENTIONS:
Drug: levosimendan — Participants randomized to to the intervention will receive levosimendan. The infusion is administered over 24 hours, starting at a dose of 0.1 µg/kg/min. After 4 hours, the dose may be increased to 0.2 µg/kg/min if tolerated, based on clinical judgment. A maximum of four treatment cycles may be given if the patient is not successfully weaned from mechanical ventilation within 7 days.
  Arms: Intervention group
Drug: Soluvit — Participants randomized to this arm will receive a placebo consisting of Soluvit diluted in glucose 5%, administered as an intravenous infusion over 24 hours. The infusion will mimic the Levosimendan administration protocol, starting at 0.1 µg/kg/min and potentially increasing to 0.2 µg/kg/min after 4 hours, to maintain blinding. A maximum of four placebo treatment cycles may be administered if the patient is not successfully weaned from mechanical ventilation within 7 days.
  Arms: Control group
Other: Standard care — All patients in this arm will receive standard ICU care, including daily assessments for readiness to wean from invasive ventilation.

SUMMARY:
Prolonged weaning from mechanical ventilation is a common and serious challenge in the ICU, associated with increased morbidity, mortality, and length of stay. Diaphragm dysfunction plays a key role in weaning failure, and current strategies to support respiratory muscle function are limited. Levosimendan is a calcium sensitizer that enhances cardiac and skeletal muscle contractility, including the diaphragm, without increasing oxygen demand.

The investigators hypothesize that treatment with Levosimendan in difficult-to-wean ICU patients will improve diaphragm function and thereby shorten the duration of mechanical ventilation compared to placebo.

DETAILED DESCRIPTION:
Objective: To assess the effect of levosimendan on the number of ventilator-free days up until day 28.

Study design: WEANLESS is an investigator-initiated, multicenter, double blind, randomized clinical superiority trial in ventilated adult patients admitted to the ICUs of participating hospitals.

Study population: This study will include 250 patients who are invasively ventilated for more than 48 hours and failed at least one SBT. Patients are enrolled from participating ICUs and randomized within 24 hours after failing their first SBT.

Intervention:

Patients will be randomly assigned in a double-blind manner to receive either levosimendan or placebo. The study medication will be administered as a continuous intravenous infusion over 24 hours, starting at a dose of 0.1 µg/kg/min, with the option to increase to 0.2 µg/kg/min after 4 hours if well tolerated. If weaning is not successful after 7 days, a maximum of four treatment cycles may be given. All patients will continue to receive standard ICU care, including daily assessments of readiness to wean from mechanical ventilation.

In addition to the intervention, health-related quality of life will be assessed using the EQ-5D-5L questionnaire at baseline, 3 months, and 12 months after inclusion. Dyspnea scores will be recorded daily after extubation until ICU discharge.

Main study parameters/endpoints: The primary endpoint of the study is the number of ventilator-free days and alive (VFD) at day 28 from randomization. This is a composite endpoint combining both mortality and the duration of ventilation. Secondary outcomes include ventilator-free days at day 90, dyspnea scores, reintubation rates, ICU readmission, ICU length of stay, hospital length of stay and mortality. Safety outcomes include the occurrence of cardiac arrhythmias, changes in vasopressor requirements and other adverse events related to levosimendan.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The burden for participants is minimal. Levosimendan is a registered drug with a known safety profile and is already used in critical care settings. The placebo is an infusion with Soluvit. All other care follows standard ICU procedures. Data will be collected from the electronic medical record and routine monitoring. No additional invasive procedures are required solely for the main study.

ELIGIBILITY:
Inclusion Criteria:

* Invasively ventilated > 48 hours.
* Failed at least one spontaneous breathing trial (SBT).
* Age above 18 years.
* Female patients with age < 60 must have a negative pregnancy test (blood or urine) prior to participation.

Exclusion Criteria:

* Pre-existing neuromuscular disease (congenital or acquired)
* Endotracheally intubated primarily for neurological reason (e.g., traumatic brain injury, intracranial haemorrhage, epilepsy, intracranial infection), or developed severe intracranial haemorrhage/infarction during ICU stay.
* Contra-indications for levosimendan: severe renal failure (creatinine clearance <30mL/min) unless managed with appropriate continuous kidney replacement therapy (such as CRRT), severe liver failure (Child-Pugh class C), history of torsade des pointes; known significant mechanical obstructions affecting ventricular filling/ outflow or both; prolonged QTc interval (QTc > 470ms); breast feeding; known hypersensitivity to levosimendan.
* Treatment with intermittent haemodialysis.
* Treatment limitation decision in place: do not reintubate
* Previous treatment with levosimendan within 30 days.
* Currently in another interventional trial that might interact with study drug or primary outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the number of ventilator-free days and alive (VFD) at day 28 from randomization. This is a composite endpoint combining both mortality and the duration of ventilation. | From randomization up until day 28.
  In case of death, the subject will be assigned a value of 0 VFD. Day 0 will be defined as the day of randomization.

SECONDARY OUTCOMES:
The number of ventilator-free days from randomization up until day 90. | From randomization up until day 90.
The number of days from randomization to successful weaning from invasive ventilation. | From randomization up until day 90.
  Weaning success defined as: for intubated patients extubation without death or reintubation within the next 7 days, or discharge from the ICU without invasive ventilation within 7 days. Whichever comes first.
  For tracheostomized patients, weaning success is defined as ventilation through tracheostomy without any invasive ventilation during 7 consecutive days, or discharged from the ICU with unassisted breathing, whichever came first.
ICU mortality | From randomization up until day 28.
ICU mortality | From randomization up until day 90.
Dyspnea sensation | From extubation up until day 28 or ICU discharge whichever comes first.
  Dyspnea will be assessed daily at the end of the spontaneous breathing trial using the Visual Analogue Scale (VAS). This is a scale from 0 to 10, where 0 means no dyspnea sensation at all and 10 the worst you have ever experiences. After extubation, dyspnea scores will be recorded daily in the morning until ICU discharge. Dyspnea sensation will be quantified as the median score from the first to the last measurement and a difference of ≥1 point on the VAS will be considered clinically meaningful.
Quality of life at baseline and at follow up after 3 and 12 months. | From randomization up until 3 and 12 months.
  The EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire will be used to assess health-related quality of life at baseline, and again at 3 and 12 months after randomization. Higher scores indicates better health status.
The number of patients with a reintubation (for endotracheally intubated patients) or reinstitution of invasive ventilation (for tracheostomized patients) within 7 days after liberation. | From randomization up until day 90.
  An endotracheal intubation beyond 7 days is not considered a "reintubation" but will be classified as a new event.
ICU readmission within 90 days. | From randomization up until day 90.
The number of days with non-invasive respiratory support (high flow nasal canula or non-invasive ventilation). | From randomization up until day 28.
The length of stay in the ICU. | From randomization up until day 90.
The length of stay in the hospital. | From randomization up until day 90.
Plasma concentration of levosimendan | From 24 hours after start of the first dose of medication up until 120 hours after start of the fist dose of medication.
  Blood samples will be collected at predefined time points ( after 24 hours, 48 hours, 72 hours and 120 hours) to determine the plasma concentration of levosimendan following intravenous administration.
Incidence of clinically significant blood pressure change | From randomization until day 28 or ICU discharge whichever comes first.
  Number of participants with a deviation of ≥20% from baseline mean arterial pressure (MAP), sustained for at least 10 minutes, as monitored continuously during infusion as part of routine ICU care.
Incidence of clinically significant heart rate change | From randomization until day 28 or ICU discharge whichever comes first.
  Number of participants with a deviation of ≥20% from baseline heart rate, sustained for at least 10 minutes, as monitored continuously during infusion as part of routine ICU care.
Vasopressor and inotropic durg use during ICU stay | From randomization until ICU discharge or day 28 whichever comes first.
  Use of vasopressors and/or inotropic drugs will be recorded daily from the start of study medication until ICU discharge. Data collected will include the generic drug name and daily dose.
Incidence and type of cardiac dysrhythmia detected by continuous ECG monitoring | From start of infusion up to 30 hours after initiation
  Continuous ECG monitoring will be used to detect cardiac dysrhythmias up to 30 hours after initiation of study medication. Detected dysrhythmias will be categorized by type.
Daily fluid balance | From randomization up until day 28 or discharge on the ICU, whichever comes first.
  Daily assessment of the fluidbalance

CONTACTS AND LOCATIONS:
Locations (8):
- Netherlands (8):
  - Rijnstate Ziekenhuis Stichting, Arnhem, Gelderland
  - Intensive Care Medicine, Radboud University, Nijmegen, Gelderland
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Jeroen Bosch Ziekenhuis Stichting, 's-Hertogenbosch, North Brabant
  - Catharina Ziekenhuis Stichting, Eindhoven, North Brabant
  - Erasmus Universitair Medisch Centrum Rotterdam (Erasmus MC), Rotterdam, South Holland
  - Sint Franciscus Vlietland Groep Stichting, Rotterdam, South Holland
  - Maasstad Ziekenhuis Stichting, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided